CLINICAL TRIAL: NCT03857191
Title: Nutritional and Psychocomportemental Reeducation, Sleep Apnea and Comorbidities in Overweight and Obese Subjects
Brief Title: Nutritional Rehabilitation and Sleep Apnea in the Obese
Acronym: DIETSLEEP
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Groupe Éthique et Santé (Industry)
Responsible Party: Sponsor
Other Study IDs: 38RC18.267; 2018-A02617-48 (Other: ID RCB)
Record Dates: First submitted 2019-02-20; First posted 2019-02-27 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Obese; Sleep Apnea, Obstructive
Keywords: obesity; sleep apnea; hypertension; type 2 diabetes; CPAP
MeSH Terms: conditions — Obesity; Sleep Apnea, Obstructive; Sleep Apnea Syndromes; Hypertension; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients already treated for OSA: The first group involves patients already diagnosed and treated for sleep apnea that will follow the nutritional psychocomportemental rehabilitation
  Interventions: Dietary Supplement: Nutritional psychocomportemental rehabilitation
- Patients with a high OSA risk: This group concerns patients with a high OSA risk according to their Berlin questionnaire score that will follow the nutritional psychocomportemental rehabilitation
  Interventions: Dietary Supplement: Nutritional psychocomportemental rehabilitation
- Patients with a low OSA risk: This group concerns patients with a low OSA risk according to their Berlin questionnaire score that will follow the nutritional psychocomportemental rehabilitation
  Interventions: Dietary Supplement: Nutritional psychocomportemental rehabilitation

INTERVENTIONS:
Dietary Supplement: Nutritional psychocomportemental rehabilitation — Nutritional psychocomportemental rehabilitation

SUMMARY:
In obese patients, the prevalence of obstructive sleep apnea (OSA) is around 40% in men and 30% in women. Weight loss after bariatric surgery significantly improves OSA, with 75% of patients having a reduction in OSA severity or becoming non-apneic. We hypothesize a similar effect on OSA of nutritional and psychocomportemental rehabilitation for obese patients. However, we expect weight loss and blood pressure reduction to probably be lower in obese patients who have OSA and nutritional rehabilitation alone than in those who are treated for their OSA or are without OSA. To address this question, we will conduct an observational study on obese patients, treated or not for OSA, following nutritional and psychocomportemental rehabilitation.

DETAILED DESCRIPTION:
In obese patients, OSA prevalence is around 40% in men and 30% in women. Being overweight or obese are independent risk factors for OSA, and the prevalence increases with body mass index (BMI). Weight loss after bariatric surgery is one treatment for OSA, 75% of patients having a reduction in OSA severity or becoming non-apneic. OSA and obesity both induce type 2 diabetes, hypertension and/or nonalcoholic fatty liver disease (NAFLD). A randomized study (Chirinos et al. NEJM 2014) demonstrated a better improvement in blood pressure, triglyceride levels or insulin resistance with weight loss alone or weight loss associated with continuous positive airway pressure (CPAP) than with CPAP alone. We hypothesize a similar effect of nutritional and psychocomportemental rehabilitation on OSA. However, weight loss and blood pressure improvements could be lesser in untreated OSA patients than in treated OSA or non-OSA patients. It has been demonstrated that bariatric surgery reduces medication use such as antihypertensive or antidiabetic drugs, and thus a secondary objective is to determine whether nutritional and psychocomportemental rehabilitation similarly reduces medication use by the overweight and obese.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 25 kg/m² and/or waist circumference > 80 cm in women or 94 cm in men
* Patients registered to follow a nutritional psychocomportemental reeducation program with the "Ethique et Santé" group

Exclusion Criteria:

- Subjects covered by articles L1121-5 to L1121-8 of French law

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Overweight and obese patients
Sampling Method: Non-Probability Sample
Enrollment: 396 (Actual)
Dates: Start 2019-03-22 (Actual); Primary Completion 2022-04-11 (Actual); Study Completion 2022-05-16 (Actual)

PRIMARY OUTCOMES:
Difference in OSA risk before and after nutritional and psychocomportemental rehabilitation | 25 weeks
  Berlin questionnaire score of patients will be compared before and after weight loss (if any) by nutritional psychocomportemental reeducation

SECONDARY OUTCOMES:
Difference in daytime sleepiness before and after nutritional and psychocomportemental rehabilitation | 25 weeks
  Epworth sleepiness score of patients will be compared before and after weight loss by nutritional psychocomportemental rehabilitation
Weight loss according to OSA status | 25 weeks
  Weight loss will be compared according to the somnolence and/or OSA risk defined by Berlin score
Change in Blood pressure according to OSA status | 25 weeks
  Blood pressure reduction between the beginning and the end of the dietary program will be compared according to OSA risk defined by Berlin score
Change in Medication use according to OSA status | 25 weeks
  Change in the number of antihypertensive, antidiabetic and lipid lowering drug use will be compared according to the change in Berlin questionnaire score
To assess the effect of Weight loss on OSA | 25 weeks
  To determine the percentage of patients stopping CPAP treatment after weight loss

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Louis PEPIN, MD, PhD, Principal Investigator — Grenoble Alpes University Hospital
Locations (1):
- Chu Grenoble Alpes, Grenoble, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Bailly S, Fabre O, Cals-Maurette M, Pantagis L, Terrail R, Legrand R, Astrup A, Pepin JL. Impact of a Weight-Loss Rehabilitation Program on Sleep Apnea Risk and Subjective Sleepiness in Patients with Overweight/Obesity: The DietSleep Study. J Clin Med. 2022 Nov 22;11(23):6890. doi: 10.3390/jcm11236890. PMID 36498465